CLINICAL TRIAL: NCT00851981
Title: Effect of Oral S-Adenosylmethionine Administration on Abnormalities of Hepatic Methionine Metabolism and Disease Progression in Alcoholic Liver Disease. A Randomized, Double Blind, Placebo-controlled Trial
Brief Title: Randomized, Controlled Trial of S-adenosylmethionine in Alcoholic Liver Disease
Acronym: RCT SAMe
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Loma Linda University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Michel H. Mendler, M.D. / PI, Loma Linda Univeristy
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 55302; 1R21AA014269-01A1 (NIH)
Record Dates: First submitted 2009-02-24; First posted 2009-02-26 (Estimated); Last update posted 2010-09-13 (Estimated); Status verified 2010-09

CONDITIONS: Alcoholic Hepatitis
Keywords: Alcohol Liver Disease
MeSH Terms: conditions — Hepatitis, Alcoholic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator)
  Interventions: Other: Placebo
- SAMe (Active Comparator)
  Interventions: Dietary Supplement: SAMe

INTERVENTIONS:
Other: Placebo — TID
  Arms: 1
Dietary Supplement: SAMe — 300 mg TID
  Arms: SAMe

SUMMARY:
Background: Alcoholic liver disease is one of the most important causes of chronic liver disease in this country. There is currently no treatment for chronic alcoholic liver disease other than abstinence. Hepatic methionine metabolism is abnormal in these patients and one of the consequences is depletion of S-adenosylmethionine (SAMe) levels, which can affect numerous important cellular processes. SAMe has been increasingly utilized for the treatment of liver diseases although the protective mechanisms remain unclear. A recent randomized double-blind trial using SAMe in patients with alcoholic liver disease and found improvement in 2-year survival in those with less advanced liver disease. However, important changes in methionine metabolism and histological changes were not included in the study. Aim: The goal of this study is to determine the effect of SAMe administration on key metabolic abnormalities of the methionine cycle and on the recovery from alcoholic liver disease.

DETAILED DESCRIPTION:
Methods: This is a randomized, double blind, placebo-controlled trial. Thirty patients with stable alcoholic hepatitis (Maddrey Score < 32) without cirrhosis who meet entry criteria will receive either 400 mg of SAMe (n=15) or placebo (n=15) three times a day for the duration of one year. History, physical assessment, various blood tests and a liver biopsy will be performed prior to treatment. Patients will have repeat blood tests on subsequent follow-up visits every month for the first two months, then every two months thereafter. They will also be encouraged to abstain from alcohol during these visits. A post-treatment liver biopsy will be obtained at the end of the trial. The primary outcome parameters include serum homocysteine, SAMe and TNFalpha levels, and the expression of key hepatic enzymes of the methionine cycle and of hepatic SAMe and glutathione levels. Histological progression of alcoholic liver disease, clinical and biochemical indices of liver disease, and quality of life assessment will also be examined.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be chronic alcohol users, defined by a history of ethanol consumption on average > 40g/day for women and 60g/day for men for at least 1 year before inclusion.
* The presumptive diagnosis for alcoholic hepatitis will be: recent binge drinking; compatible physical findings (one or more: jaundice, enlarged liver, hepatic bruit, abdominal pain, loss of appetite, nausea); and a compatible biochemical profile (moderate elevation of AST over ALT, elevated total serum bilirubin); or a liver-spleen colloid scan suggestive of reticulo-endothelial redistribution and hepatic arterialization.
* The diagnosis of alcoholic hepatitis must be confirmed on liver biopsy, showing typical features of acute sclerosing hyaline necrosis 70.
* The degree of portal fibrosis as determined on liver biopsy, graded according to the Knodell score-modified by Ishak 71 must be less than or equal to 5 out of a possible score of 6, 6 indicating cirrhosis.
* The alcoholic hepatitis must be "stable", i.e. not requiring treatment by either pentoxifylline 72 or prednisone, with a Maddrey Score 73 {(PTpatient - PTcontrol) x 4.6 + TBmg/dL} < 32.
* Patients must be willing to participate in the trial, remain abstinent to alcohol, and compliant to the treatment regimen, and undergo a post-treatment liver biopsy.

Exclusion Criteria:

* Patients who have either compensated cirrhosis (biopsy proven) or a clinical picture of severe cirrhosis defined as Child's class C and/or with a recent history (within one month) of decompensated liver disease (history of ascites, encephalopathy or variceal bleeding within one month of trial entry). These patients have reduced life expectancy below one year and are most often severely coagulopathic and cannot be biopsied.
* Patients who have severe acute alcoholic hepatitis of poor prognosis defined as a Maddrey Score > 32. These patients have a mortality rate of 50% during their hospitalization period when untreated by either prednisone or pentoxifylline.
* Patients who are receiving hepatotropic treatments such as colchicine, penicillamine, corticosteroids, ursodeoxycholic acid, and pentoxifylline.
* Patients who are receiving known hepatotoxic long-term treatments such as NSAIDs, statins, neuroleptics, certain anti-convulsive medications, or high-dose acetaminophen.
* Patients suspected of having hepatocellular carcinoma.
* Patients who have contra-indications to liver biopsy.
* Patients who have a liver biopsy that does not yield sufficient specimen for analyses.
* Patients who have untreated deficiencies of folic acid, vitamin B6 or B12.
* Patients who have chronic active Hepatitis B or C, hemochromatosis, autoimmune hepatitis, or a cholangiopathy.
* Patients with psychotic disorders, and in particular manic depression (contra indication to SAMe treatment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-10; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Change in plasma homocysteine, hepatic GSH and SAMe levels and hepatic expression of TNF,MAT1A,MAT2A,MS,CBS and BHMT. | 1 year

SECONDARY OUTCOMES:
Changes in routine liver pathology,c-myc expression and markers of apoptosis, stellate cell activation and hepatocyte proliferation. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Michel H Mendler, M.D., Principal Investigator — Loma Linda Univeristy
Locations (1):
- Loma Linda University, Loma Linda, California, United States